CLINICAL TRIAL: NCT03794687
Title: The Distal (SnUffbox) Radial artERy Access for Coronary Angiography and Interventions (SUPER-Prospective)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201802924
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Coronary Angiography
Keywords: Left heart catheterizations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Distal Radial Artery: Left heart catheterization via the distal radial artery (dorsal aspect of the hand at the base of the thumb).
  Interventions: Procedure: Left heart catheterization

INTERVENTIONS:
Procedure: Left heart catheterization — Catheterization via the distal radial artery

SUMMARY:
The study team aims to perform a prospective observational case series of one hundred consecutive distal radial artery heart catheterizations to evaluate the safety and feasibility of distal radial access. Distal radial artery access has evolved in the past few years as an alternative to the standard radial artery access for coronary angiography and interventions. However, the available data on the distal radial artery access for coronary angiography and interventions is limited to case reports and small retrospective case series. To date, no prospective randomized data is available. Therefore, the investigators aim to perform a prospective observational case series of one hundred sequential left heart catheterizations performed via distal radial artery to evaluate the safety and feasibility of the distal radial artery access.

DETAILED DESCRIPTION:
Despite the abundance of data supporting the use of the radial artery compared to the femoral artery, data on the use the distal radial access site in the anatomical snuffbox is limited. Most of the available literature on the distal radial access comes from case reports and small retrospective case series looking primarily at the feasibility and success rates with this approach (4-6). Crossover rate from proximal radial to femoral approach in a prior randomized controlled trial was reported at 3.7% (2). A similar rate has been reported in case series studies of distal radial access, with success rates ranging from 88.6% to 96.3% (4-6). No cases of radial artery occlusion, hematoma, or hand paresthesia were reported in any of these series. Given the promising results with the distal radial approach, its use has expanded to many cardiac catheterization laboratories across the country. However, prospective randomized data comparing distal versus the conventional proximal radial arterial access sites is warranted.

Therefore, the aim of this study is to compile a prospective observational case series to evaluate the safety and feasibility of distal radial artery access in a prospective case series. If an acceptable safety profile can be demonstrated, the case series will be followed with a randomized controlled trial directly comparing distal to standard proximal radial artery approach.

Specific Aims and study hypothesis:

The primary aim of the present study is to assess the safety and feasibility of distal radial arterial access. The study hypothesis is that distal radial access for coronary angiography is associated with similar incidence rates of access site related complications compared to complication rates previously reported with the standard proximal radial artery access.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo diagnostic left heart catheterization with or without percutaneous coronary intervention.

Exclusion Criteria:

* Hemodynamically unstable (on vasopressor continuous infusion, on mechanical support) patients.
* Patients undergoing emergent left heart catheterization for ST-elevation myocardial infarction.
* Full oral anticoagulation defined as use of a direct oral anticoagulant (DOAC) within 24 hours or an INR over 2.0 the day of the procedure.
* Active bleeding or known history of blood dyscrasia or bleeding diathesis.
* History of ipsilateral arteriovenous fistula or vascular surgical intervention.
* Patients unable to undergo distal radial artery access due to anatomical deformities, limited mobility, or other.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of up to one hundred consecutive patients undergoing left heart catheterization via the distal radial artery (dorsal aspect of the hand at the base of the thumb) will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Safety of distal radial arterial access | 10 Minutes
  Incidence of any radial access complication defined as the composite of radial artery occlusion, radial artery vasospasm, other access site related bleeding or vascular complications, or hand dysfunction

SECONDARY OUTCOMES:
Feasibility of distal radial arterial access defined as failure of access within 10 minutes with conversion to an alternative arterial access site. | 10 Minutes
  Failure of access will be defined as inability to obtain access within 10 minutes from initial administration of local anesthetic to successful cannulation of the radial artery.
Patient satisfaction | 30 Minutes
  Patient satisfaction will be assessed with a patient satisfaction survey following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andres Pineda Maldonado, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States